CLINICAL TRIAL: NCT04005339
Title: NAPOLI-2: Phase II Study of Fluorouracil, Leucovorin, and Nanoliposomal Irinotecan in Previously Treated Advanced Biliary Tract Cancer
Brief Title: NAPOLI-2: Fluorouracil, Leucovorin, and Nanoliposomal Irinotecan in Biliary Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0877
Record Dates: First submitted 2019-06-27; First posted 2019-07-02 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Advanced Biliary Tract Cancer
Keywords: Advanced Biliary Tract Cancer; Biliary Tract Cancer; GI Cancer; Biliary Cancer; NAPOLI-2
MeSH Terms: conditions — Biliary Tract Neoplasms; Gastrointestinal Neoplasms | interventions — irinotecan sucrosofate; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Nanoliposomal irinotecan 70 mg/ IV over 90 minutes, every 14 days. Leucovorin 400 mg/ IV over 30 minutes, every 14 days. Fluorouracil 2,400 mg/m IV over 46 hours.
  Interventions: Drug: Nanoliposomal Irinotecan; Drug: Leucovorin; Drug: Fluorouracil

INTERVENTIONS:
Drug: Nanoliposomal Irinotecan — Nanoliposomal irinotecan 70 mg/ IV over 90 minutes, every 14 days
Drug: Leucovorin — Leucovorin 400 mg/ IV over 30 minutes, every 14 days.
Drug: Fluorouracil — Fluorouracil 2,400 mg/m IV over 46 hours.

SUMMARY:
This is a study to evaluate the clinical activity of the combination of fluorouracil, leucovorin, and nanoliposomal irinotecan as second-line treatment in patients with advanced biliary tract cancers following gemcitabine and platinum chemotherapy.

DETAILED DESCRIPTION:
This is a single arm, open label, multicenter phase II study to evaluate the clinical activity of the combination of fluorouracil, leucovorin, and nanoliposomal irinotecan as second-line treatment in patients with advanced biliary tract cancers following gemcitabine and platinum chemotherapy. Patients with advanced biliary tract cancers who have adequate performance status and adequate hepatic and renal function will be eligible. Patients may have received adjuvant chemotherapy and/or radiation therapy prior to enrolling in the trial, but a minimum of 6 months between adjuvant chemotherapy and this current therapy are required. Patients may continue on study as long as they are tolerating treatment and do not have progression of disease by RECIST v1.1 criteria. Response assessments will occur using imaging (CT or MRI) every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically-confirmed biliary tract cancer (cholangiocarcinoma or gallbladder adenocarcinoma), unresectable or metastatic
* Disease progression on or intolerance of gemcitabine- and platinum-based chemotherapy
* No more than 1 prior line of chemotherapy for unresectable or metastatic disease (adjuvant therapy does not count)
* Measurable disease by RECIST v1.1 criteria
* ECOG performance status of 0-1
* At least 18 years of age
* HIV-positive patients are eligible provided: Stable HAART regimen, No concurrent prophylactic antibiotics or antifungals, and CD4 count above 250 and undetectable viral load
* Adequate bone marrow, hepatic, and renal function
* Consent to access archived tumor tissue if available (available tissue is not required for enrollment)

Exclusion Criteria:

* Ampullary adenocarcinoma
* Woman who are pregnant or breastfeeding
* Anti-cancer treatment within 3 weeks prior to enrollment
* Prior irinotecan or nanoliposomal irinotecan
* Central nervous system metastases unless stable for at least 4 weeks and at least 2 weeks off corticosteroids
* Exposure to a strong CYP3A4 inducer, strong CYP3A4 inhibitor, or strong UGT1A1 inhibitor within 2 weeks of study start
* Known concurrent malignancy or other malignancy within 3 years except for non-melanomatous skin cancers, prostate or cervical cancers following curative therapy, or superficial bladder cancer
* Bowel obstruction
* Allergy or hypersensitivity to fluoropyrimidines, irinotecan, or nanoliposomal irinotecan
* Clinically significant liver disease: Patients with resolved hepatitis B infection are eligible if HBsAg testing is negative; Patients with resolved hepatitis C infection are eligible if viral RNA PCR is negative
* Severe infections within 4 weeks prior to enrollment
* Major surgery within 4 weeks prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The efficacy of fluorouracil, leucovorin, and nanoliposomal irinotecan in advanced biliary tract cancers following progression on or intolerance of gemcitabine and platinum chemotherapy. | 4 months
  Defined as positive if there is no evidence of disease progression (PD) at 4 months, as measured by RECIST v1.1 criteria

SECONDARY OUTCOMES:
Overall response rate (ORR). | 6 months
  The activity of fluorouracil, leucovorin, and nanoliposomal irinotecan in patients with advanced biliary tract cancers treated following progression on or intolerance of gemcitabine and platinum chemotherapy measured in terms of best overall response rate (ORR).
Median progression-free survival (mPFS). | 6 months
  The activity of fluorouracil, leucovorin, and nanoliposomal irinotecan in patients with advanced biliary tract cancers treated following progression on or intolerance of gemcitabine and platinum chemotherapy measured in terms of median progression-free survival (mPFS).
Median overall survival (mOS). | 6 months
  The activity of fluorouracil, leucovorin, and nanoliposomal irinotecan in patients with advanced biliary tract cancers treated following progression on or intolerance of gemcitabine and platinum chemotherapy measured in terms of median overall survival (mOS).
Median time to disease progression (mTTP). | 6 months
  The activity of fluorouracil, leucovorin, and nanoliposomal irinotecan in patients with advanced biliary tract cancers treated following progression on or intolerance of gemcitabine and platinum chemotherapy measured in terms of median time to disease progression (mTTP).
Disease control rate (DCR). | 6 months
  The activity of fluorouracil, leucovorin, and nanoliposomal irinotecan in patients with advanced biliary tract cancers treated following progression on or intolerance of gemcitabine and platinum chemotherapy measured in terms of disease control rate (DCR).
Median duration of disease control (DDC). | 6 months
  The activity of fluorouracil, leucovorin, and nanoliposomal irinotecan in patients with advanced biliary tract cancers treated following progression on or intolerance of gemcitabine and platinum chemotherapy measured in terms of median duration of disease control (DDC).
Maximum change in tumor marker, CA19-9. | 6 months
  The activity of fluorouracil, leucovorin, and nanoliposomal irinotecan in patients with advanced biliary tract cancers treated following progression on or intolerance of gemcitabine and platinum chemotherapy measured in terms of maximum change in tumor marker, CA19-9.

OTHER OUTCOMES:
Blood for the analysis of circulating tumor DNA as a surrogate marker of disease burden. | 6 months
  Correlation of dynamics of circulating tumor DNA change compared with change in CA19-9.
Archived tumor tissue using next-generation sequencing (NGS) and immunohistochemistry (IHC) in order to elucidate potential mutational biomarkers predictive of response to fluorouracil, leucovorin, and nanoliposomal irinotecan. | 6 months
  Correlation of tumor genetic mutations and protein expression levels with progression-free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Weinberg, MD, Study Chair — Georgetown University
Locations (4):
- United States (4):
  - Lombardi Comprehensive Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Washington University School of Medicine- Siteman Cancer Center, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No